CLINICAL TRIAL: NCT05545033
Title: Evaluating the Feasibility and Acceptability of the Use of Virtual Reality in Pain Management in Hospitalized Patients
Brief Title: Use of Virtual Reality in Pain Management in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Lydia Li Weiling, Consultant, Department of Anaesthesia and Surgical Intensive Care, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIRTUAL01
Record Dates: First submitted 2022-09-11; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pain, Acute; Pain, Chronic
Keywords: virtual reality; pain management; inpatients
MeSH Terms: conditions — Acute Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Open-label, single centre, single-arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality intervention (Experimental): Comparison of pain and anxiety levels before and after VR intervention within the same patient.
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — 5 to 15 minutes of virtual reality exposure

SUMMARY:
Acute and chronic non-cancer pain is a common healthcare problem locally and globally, leading to many inpatient admissions for poorly controlled pain. The World Health Organisation has declared that access to adequate pain control is a fundamental human right. Yet in our current practice, both acute and chronic non-cancer pain remain poorly controlled.

There is passive over-reliance on pharmacological agents and interventional procedures in the management of pain. The opioid epidemic with issues of dependence, misuse, and overdose is especially concerning. Therefore, there is a pertinent clinical need to find sustainable non-pharmacological adjuncts in the complex management of pain.

Virtual reality (VR) involves the use of technology to create a three-dimensional multisensory artificial environment replacing real-world sensory inputs. Initially created solely for entertainment purposes, VR applications have since expanded and made its way into healthcare. In Pain Medicine, the application of VR has been promising. There is currently no VR study done in our local population who suffer from pain issues. In our study, we aim to test the feasibility of applying the use of VR in patients admitted inpatient due to pain issues. We believe that VR can be used as an adjunctive tool improve pain management and patient satisfaction.

DETAILED DESCRIPTION:
Patients who agree to participate in the study will undergo the following procedures:

1. Provide written informed consent,
2. Provide baseline demographic information,
3. Provide baseline pain and anxiety ratings,
4. Undergo 5 to 15 minutes VR exposure,
5. Take 3 to 5 minutes break,
6. Undergo 5 to 15 minutes VR exposure,
7. Provide post-intervention pain and anxiety ratings,
8. Complete validated questionnaires.

The Oculus Go Head-Mounted Devices (HMD) will be put in place on the patients as follows:

1. Patient places sanitary hairnet on head,
2. Patient places disposable face liners secured by rubber bands over their ears,
3. Study coordinator places pre-sanitized Oculus Go HMD over patient's disposable face mask and adjusts straps for comfort.

Trial Product:

This study will be using immersive VR technology for intervention and management of acute and chronic pain. It will deploy the latest commercially available all-in-one HMDs as an adjunct to pain management in an inpatient hospital setting.

The VR hardware configuration and all content is currently being developed by technology partner Vue Networks, a leader in the development of VR content for implementation in education and training for the Social Sciences sector and in health and mental wellness for community and institutional usage, such as for the elderly and demented in hospitals and in nursing homes. Content experts consulted include certified MBCT practitioners as well as VR content researchers in Singapore and Germany.

VR Hardware: This study will utilize the Oculus Go all-in-one HMD set designed by Facebook Reality Labs. This is the first wireless HMD created that is able to display 4K images in a 3-degrees of Freedom environment.

VR Software: In immersive VR, high resolution (minimum 4K) 360-degree video and 3D computer graphics and paired with suitable ambience sounds and audio cues to fully immerse the user in the selected environment.

The proposed VR experiences include the following:

1. Gardens by the Bay - Limit-Oriented Therapy (Cognitive Restructuring)
2. Animated Nature Environment - Enhance-Oriented Therapy (Mindfulness Meditation)
3. Animated Beach Environment - Active-Oriented Therapy (Behavioural Activation)
4. Underwater Fish & Mammals - Integrated Treatment (Multimodal Treatment)

Content will be a mixture of life-action and animation, as well as foreign and local

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalised patients with complain of pain issues (at least one of the following),

   * Acute pain
   * Acute exacerbations of chronic pain
   * Chronic non-cancer pain
   * Post-procedural pain (limited to those who undergo procedures with < 2 hours in duration)
2. Age equal or more than ≥ 21 years,
3. No visual or hearing impairment,
4. English literacy.

Exclusion Criteria:

1. Cancer-related pain,
2. Comorbidities affecting usage of VR e.g. motion sickness, stroke, seizure, dementia, transmissible diseases, severe facial eczema,
3. Undergoing litigation.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Patient acceptability and tolerability | post-intervention (up to 1 hr)
  Validated questionnaires - patient experience satisfaction (0 to 10; 0-worst outcome, 10-best outcome), System Usability Scale (<50-not acceptable, 50-70-marginal, >70-acceptable)

SECONDARY OUTCOMES:
Clinical efficacy of virtual reality | pre- and post-intervention (up to 1hr)
  Pain and anxiety scores (0 to 10; 0-best outcome, 10-worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Li, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mosadeghi S, Reid MW, Martinez B, Rosen BT, Spiegel BM. Feasibility of an Immersive Virtual Reality Intervention for Hospitalized Patients: An Observational Cohort Study. JMIR Ment Health. 2016 Jun 27;3(2):e28. doi: 10.2196/mental.5801. PMID 27349654
- [Background] Jones T, Moore T, Choo J. The Impact of Virtual Reality on Chronic Pain. PLoS One. 2016 Dec 20;11(12):e0167523. doi: 10.1371/journal.pone.0167523. eCollection 2016. PMID 27997539